CLINICAL TRIAL: NCT04463693
Title: Pilot Study of Etonogestrel Contraceptive Implant Insertion at an Alternative Subdermal Scapular Site
Brief Title: Shoulder Contraceptive Implant Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20-0574
Record Dates: First submitted 2020-07-01; First posted 2020-07-09 (Actual); Results first posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-05

CONDITIONS: Contraception
MeSH Terms: interventions — etonogestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Insertion of the etonogestrel contraceptive implant subdermally over the non-dominant scapula
  Interventions: Drug: Etonogestrel implant

INTERVENTIONS:
Drug: Etonogestrel implant — Insertion of the contraceptive implant at an alternative insertion site located over the scapula

SUMMARY:
This study will be the first to establish pharmacokinetic curves for the etonogestrel contraceptive implant with scapular subdermal insertion. By obtaining this pharmacokinetic data, the investigators can compare this data to already published pharmacokinetic data with conventional implant insertion. This comparison can provide some reassurance that the absorption and distribution of etonogestrel from the contraceptive implant with scapular insertion is similar to that found with conventional insertion. With similar pharmacokinetic properties, the investigators would expect scapular insertion of the implant to maintain similar contraceptive efficacy for the populations of women that may benefit from this alternative insertion site. Preliminary safety data will also enrich the understanding of any potential insertion site side effects with subdermal scapular implant insertion, as the investigators currently only have a single case report with side effect outcomes. The investigators can then use this pilot data to support future larger investigations on subdermal scapular implant insertion given its complete avoidance of the neurovascular complications associated with arm insertion.

DETAILED DESCRIPTION:
The etonogestrel contraceptive implant (Nexplanon®) remains the most effective hormonal contraceptive method available in the U.S. The contraceptive implant is routinely inserted just beneath the skin on the inner-side of the non-dominant arm, but insertion at this site has resulted in rare, yet potentially morbid complications. These complications are due to the close proximity of major neurovascular structures (e.g. basilic vein, ulnar nerve) in the sulcus between the biceps and triceps muscles. Insertion of the implant deep in the arm has resulted in severe complications including migration of the implant into the pulmonary vasculature and neurological injury at the time of implant removal. Though these complications are rare, their report directly led to changes in the manufacturer's mandatory insertion training to move the implant insertion site inferiorly, though it is unlikely that this change will completely remove the risk of these rare insertion complications.

In addition to the rare complications of deep implant insertion in the arm, patients with specific medical conditions are also not ideal candidates for this standard insertion site. Patients with psychotic illnesses or development delays often require reliable contraception, but the arm insertion site for the implant is easily accessible and injuries can result from self-removal attempts among these patients. Furthermore, patients with muscular dystrophy disorders may not have adequate tissue in this region of the arm to buffer the implant from the underlying neurovascular structures. In order to address the needs of these patient populations, insertion of the contraceptive implant at an alternative subdermal scapular site has been reported in the literature. This insertion just beneath the skin overlying the inferior edge of the scapula represents an ideal alternative location for the contraceptive implant due to its location far from danger zones of neurovascular structures, inaccessibility to patients with mental illnesses, and underlying bony structure preventing unintentional deep insertion. However, more data are needed regarding the rate of drug absorption and overall safety with etonogestrel implant insertion at this alternative site.

The study will address this knowledge gap by piloting contraceptive implant insertion at this alternative scapular site among five healthy, reproductive aged women. The investigators will insert contraceptive implants at this alternative scapular site and conduct serial measurements of the amount of drug (etonogestrel) circulating in each participant's system over the course of one year. These measurements will allow us to compare the amount of circulating drug from the contraceptive implant between this alternative insertion site and the already published amounts found with standard insertion in the arm. The investigators will also ask participants about any insertion site related side effects and also general implant-related side effects (e.g. abnormal bleeding, headaches, weight gain) during the course of the study. This will provide preliminary side effect data to help us better understand patient experience with this alternative insertion site. Ultimately, the investigators hypothesize that this study will provide reassuring data that can support future larger investigations on this alternative scapular insertion site for the implant. This alternative insertion site may allow patients who otherwise are not currently candidates for the most effective hormonal contraceptive method to uptake contraceptive implants in a safe manner. This research will also allow healthcare providers to discuss an alternative site for the contraceptive implant for those patients concerned about the potential risks of deep arm insertion, thus improving patient-centered options for contraceptive implant provision.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women

Exclusion Criteria:

* Any contraindications to etonogestrel implant use based on the US Medical Eligibility Criteria for Contraceptive use (defined as class 3 or 4 recommendation)18
* Any known liver conditions that could affect drug metabolism (e.g. cirrhosis, hepatitis)
* Currently taking any medications or supplements known to be CYP3A4 inducers/inhibitors19
* Body-mass index less than 18.5kg/m2 or greater than 30kg/m2
* Currently pregnant or planning to become pregnant in the next 12 months

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Etonogestrel Implant: Insertion of the etonogestrel contraceptive implant subdermally over the non-dominant scapula
  Etonogestrel implant: Insertion of the contraceptive implant at an alternative insertion site located over the scapula
Period: Overall Study
Arm/Group | Etonogestrel Implant
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Etonogestrel Implant
Number analyzed (Participants) | 5
Age, Continuous [Median (Full Range); unit: years] | 26.0 [19.6 to 30.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5
Body mass index [Median (Full Range); unit: kg/m^2] | 25.0 [22.0 to 28.0]

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics in the Form of Serum Etonogestrel Concentrations
Description: Serum etonogestrel concentration curves measured over the first year of implant use
Time Frame: 1 week and 12 months
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Etonogestrel Implant
Number analyzed (Participants) | 5
pg/mL
  One-week post insertion | 511.7 (168.2)
  12 months post-insertion | 136.6 (21.8)

2. Secondary Outcome: Number of Participants With Side Effects
Description: Local and systematic side effects associated with etonogestrel contraceptive implant use
Time Frame: One and two weeks for "post-insertion site discomfort", over 12 months for "Amenorrhea", "Persistent bleeding", and "Intermittent bleeding"
Measure: Count of Participants; unit: Participants
Arm/Group | Etonogestrel Implant
Number analyzed (Participants) | 5
Participants
  One-week post insertion site discomfort | 4
  Two-week post insertion site discomfort | 0
  Amenorrhea | 1
  Persistent bothersome bleeding | 1
  Intermittent bleeding | 3

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Etonogestrel Implant
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 4/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etonogestrel Implant (N=5)
One week post-insertion site discomfort (Skin and subcutaneous tissue disorders) | 4 — 4 out 5 participants reported some insertion site discomfort one week after insertion of the etonogestrel implant. This is an anticipated adverse event
Persistent bothersome uterine bleeding (Reproductive system and breast disorders) | 1 — One participant reported persistent bothersome bleeding over the course of 12 months after etonogestrel implant insertion. This was an anticipated adverse event
Intermittent uterine bleeding (Reproductive system and breast disorders) | 3 — 3 out of 5 participants reported intermittent uterine bleeding over the course of 12 months after etonogestrel implant insertion. This was an anticipated adverse event

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-15): https://cdn.clinicaltrials.gov/large-docs/93/NCT04463693/Prot_SAP_000.pdf